CLINICAL TRIAL: NCT06634979
Title: Selective Lymph Node Resection for Invasive Non-small Cell Lung Cancer With the CTR of 0.5-1 and the Diameter of ≤ 2 cm: a Prospective， Single-arm, Multi-center, Phase Ⅱ Trial
Brief Title: Selective Lymph Node Resection for Invasive Non-small Cell Lung Cancer With the CTR of 0.5-1 and the Diameter of ≤ 2 cm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP-1027
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer (NSCLC); Lymph Node Dissection
Keywords: Selective lymph node dissection
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm Selective lymph node dissection (Experimental): Lower mediastinal lymph node clearance is not required for upper lobe tumors and upper mediastinal lymph node clearance is not required for lower lobe tumors in the group
  Interventions: Procedure: Selective lymph node dissection

INTERVENTIONS:
Procedure: Selective lymph node dissection — For 0.5 < CTR < 1 and ≤ 2 cm diameter cT1N0M0 invasive non-small cell lung cancer patient sex for selective lymph node (lower mediastinal lymph nodes are not required to be cleared for upper lobe tumors and upper mediastinal lymph nodes are not required to be cleared for lower lobe tumors)

SUMMARY:
The study investigated the efficacy and safety of a selective lymph node strategy (no lower mediastinal lymph node dissection for upper lobe tumors and no upper mediastinal lymph node dissection for lower lobe tumors) in patients with 0.5 < CTR < 1 and ≤ 2 cm in diameter cT1N0M0 infiltrating NSCLC, aiming to more accurately assess the prognosis of the selective lymph node dissection strategy for nodes with 0.5 < CTR < 1 and ≤ 2 cm in diameter.

DETAILED DESCRIPTION:
Selective lymph node dissection is an important idea to reduce the trauma of mediastinal lymph node dissection in early clinical patients. In a previous study, our team proposed a predictive model for mediastinal lymph node metastasis in patients with clinical T1N0 non-small cell lung cancer, and found that age, tumor size, central type, and pathologic subtype were closely related to mediastinal lymph node metastasis. In addition, our team found that adenocarcinoma in situ (AIS), minimally invasive adenocarcinoma (MIA), and invasive adenocarcinoma with predominantly adherent subtype (LPA) did not have mediastinal lymph node metastasis, and lymph node dissection was not necessary for such patients. In addition, by retrospectively studying nearly 3,000 cases of stage I-III NSCLC, we found that NSCLCs in the apical segments do not metastasize to the lower mediastinum, whereas in N1 lymph node-negative patients with negative pleural invasion, tumors in segments of the upper lobes do not metastasize to the lower mediastinal lymph nodes. On this basis, we conducted the first international prospective phase II clinical trial of a selective lymph node dissection strategy to validate the clinical feasibility of a selective lymph node dissection strategy. The main objective of this study was to develop a selective lymph node dissection strategy for cT1NOM0 invasive NSCLC with a diameter of ≤2 cm, i.e., no lower mediastinal lymph node dissection for tumors located in the upper lobe, and no upper mediastinal lymph node dissection for tumors located in the lower lobe. Further, we retrospectively analyzed 7067 NSCLC cases with systematic lymph node dissection from April 2008 to July 2022, in which the rate of mediastinal lymph node metastasis was 15.4% (1091/7067), and there was no lymph node metastasis in 209 cases of AIS/MIA/LPA, whereas in other subtypes of adenocarcinomas, the rate of mediastinal lymph node metastasis was 15.3% (106 /695). Among them, we retrospectively analyzed 360 cases of cT1N0M0 non-small cell lung cancer with 0.5 < CTR < 1.0 and found that among them, tumors located in the upper lobe had no lower mediastinal lymph node metastasis, and tumors located in the lower lobe had no metastasis in the upper mediastinal lymph nodes. For other non-small cell lung cancers with 0.5 < CTR < 1.0, if the VPI was negative, no lower mediastinal metastasis was also observed in tumors in the upper lobe and no upper mediastinal metastasis was observed in tumors in the lower lobe. In 212 cases of lung cancer not exceeding 1 cm in size, there were no lower mediastinal metastases in tumors in the upper lobe and no upper mediastinal metastases in tumors in the lower lobe.

The study investigated the efficacy and safety of a sex-selective lymph node strategy (no lower mediastinal lymph node clearance for upper lobe tumors and no upper mediastinal lymph node clearance for lower lobe tumors) in patients with 0.5 < CTR < 1 and ≤ 2 cm in diameter cT1N0M0 infiltrating NSCLC, aiming to more accurately assess the prognosis of the selective lymph node dissection strategy for nodes with 0.5 < CTR < 1 and ≤ 2 cm in diameter.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in a clinical study and be willing to follow and have the ability to complete all trial procedures;
* Age 18-80 years at time of signing informed consent (including threshold);
* ECOG score 0 or 1;
* No previous surgery for lung cancer;
* Intraoperative or postoperative pathologically confirmed non-small cell lung cancer;
* Single pulmonary nodule with mixed ground glass on CT, or multiple pulmonary nodules but the main lesion is the above nodules;
* The proportion of solid components of the nodule is between 0.5 and 1, and the total size of the nodule is less than or equal to 2 cm;
* Patients with clinical stage T1N0M0 surgically resectable;
* Primary treatment without radiotherapy or chemotherapy.

Exclusion Criteria:

* T1N0M0 with a clinical stage other than 0.5 < CTR < 1 and a diameter of ≤ 2 cm;
* Inability to perform complete surgical resection;
* cytology or histopathology confirms that it is a lung malignant tumor other than non-small cell lung cancer;
* Previous surgery for lung cancer;
* Patients who have received radiotherapy or chemotherapy for non-primary treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
2-year disease-free survival | From enrollment to the end of treatment at 2 years

SECONDARY OUTCOMES:
2-year overall survival | From enrollment to the end of treatment at 2 years

OTHER OUTCOMES:
5-year disease-free survival | From enrollment to the end of treatment at 5 years
5-year overall survival | From enrollment to the end of treatment at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No